CLINICAL TRIAL: NCT06410508
Title: Evaluation of a Brief Intervention to Improve Engagement and Recovery for At-risk Youth Enrolled in Early Intervention Services for Psychosis .
Brief Title: Evaluation of a Brief Intervention to Improve Engagement in Early Intervention Services for Psychosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Queen Elizabeth II Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Phil Tibbo, Physician, Nova Scotia Health Authority
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 62437
Record Dates: First submitted 2024-04-30; First posted 2024-05-13 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2024-05

CONDITIONS: Psychotic Disorders; Psychiatric Hospitalization; Engagement, Patient
Keywords: early phase psychosis
MeSH Terms: conditions — Psychotic Disorders; Patient Participation

STUDY DESIGN:
Intervention Model Description: Participants will not be randomized to study conditions due to recruitment difficulties and ethical concerns related to randomizing participants to a condition that has previously been demonstrated to be efficacious. Instead, participants wanting to engage in the intervention will be included in the active treatment arm and those wishing to recieve treatment as usual will be included as controls. See description of study protocol above for more detailed explanation of interventional study design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Engagement Intervention Group (experimental) (Experimental): As described in further detail in the study description: In addition to regular early intervention treatment for psychosis, participants in this group will receive a brief 2-module engagement focused psychotherapeutic orientation co-delivered by a mental health clinician and a peer support worker. This intervention will involve integration of principles of CBT and motivational interviewing in order to target previously identified affective and cognitive barriers to young adults' engagement in treatment. Treatment targets include: self-stigma, negative perceptions/beliefs towards healthcare, negative past experiences with psychiatric services, recover, and external vs internal locus of control. Participants will be guided through a standard therapeutic protocol adapted from the original Munson et al. (2022), trial targeting these barriers over 2 90-120 minute sessions delivered 1 month apart.
  Interventions: Other: Just Do You
- Treatment as Usual Group (control) (No Intervention): As described in further detail in the study description, control participants will receive the usual treatment provided at our early intervention for psychosis clinic. Treatment as usual includes psychiatric monitoring of lowest effective dose pharmaceutical treatment (e.g., antipsychotics), and various psychosocial interventions including CBT for psychosis when indicated, occupational therapy, family education and support sessions, and support for client's educational or vocational goals. Those in the engagement intervention group (experimental) will also receive this treatment in addition to the experimental engagement intervention.

INTERVENTIONS:
Other: Just Do You — As described in further detail previously, the experimental intervention is a brief psychotherapeutic intervention informed by principles of CBT and motivational interviewing that is co-delivered by a mental health clinician and peer support worker. This intervention will be a version of the initial intervention delivered in the "Just Do You" trial by Munson et al.(2022), adapted for increased suitability with our clinical population.
  Other Names: Engagement Focused Psychotherapeutic Orientation
  Arms: Engagement Intervention Group (experimental)

SUMMARY:
Negative experiences with healthcare prior to referral to early intervention services for psychosis (EIS) have been linked to poor engagement and clinical outcomes. Recent research indicates that young adults who come to EIS services thru emergency departments, urgent care, or inpatient services have significantly greater rates of future use of these services as well as more negative perceptions of EIS and diminished engagement in treatment compared to young adults referred to EIS by other pathways. These findings suggest a need for additional support to be provided to EIS patients, especially those with prior negative healthcare experiences, to maximize treatment engagement and outcomes. A recent USA-based trial of a brief intervention addressing barriers to disengagement (Just Do You), including prior negative healthcare experiences, showed promise in improving engagement and recovery. This project seeks to adapt and evaluate the Just Do You intervention to a young adult early psychosis population in Nova Scotia. The investigators aim to recruit young adults from the Nova Scotia Early Psychosis Program to engage in 2 psychotherapy/psychoeducation sessions co-led by a clinician and peer support worker. Following the intervention, the investigators will measure improvements in participants' engagement and recovery to determine the effectiveness of the program. Outcomes between participants with negative prior healthcare experiences and those without will be compared to assess differential impact of the intervention for high-risk sub-groups. This project has the potential to improve patients' engagement in EIS care and enhance recovery outcomes for young adults.

DETAILED DESCRIPTION:
Background and rationale

For young adults experiencing early phase psychosis, interactions with health services during initial help seeking are believed to be crucial in framing future attitudes towards healthcare and engagement in subsequent treatment. Young adults experiencing psychosis often encounter significant adversity during initial help-seeking. Delays to accessing suitable early intervention treatment are common, and most young adults are referred to early intervention services for psychosis (EIS) via emergency and inpatient services while experiencing acute psychosis. These referral experiences can involve law enforcement and involuntary hospitalization which are highly distressing for young adults, especially in the context of first contact with services.

In general psychiatric samples (i.e., across diagnostic groups, ages and phases of illness), prior involuntary hospitalization is associated with negative views towards subsequent treatment with views of treatment as punitive and coercive rather than therapeutic, and feelings of betrayal towards healthcare. In addition, in young adults experiencing early phase psychosis with prior hospitalization, the prevalence of PTSD diagnosis is twice that of individuals without prior hospitalization with research attributing this increased prevalence to adversity specific to individuals' prior experiences of healthcare. Individuals experiencing early phase psychosis with comorbid PTSD, often display diminished recovery and engagement in treatment. While these outcomes alone are undesirable, less is known about the relationship to between adverse experiences with healthcare and future engagement in EIS.

Recent research at the Nova Scotia Early Psychosis Program (NSEPP), has shown a relationship between referral source to EIS and subsequent health care utilization: when controlling for symptom severity and functioning, participants referred to NSEPP from urgent services (emergency, inpatient and urgent care), compared to those referred from GPs, had a greater than 3-fold use of emergency and inpatient services 2 years following their acceptance to the NSEPP. A related qualitative study further linked service users' help-seeking and referral experiences to their perceptions towards EIS and engagement in treatment; participants with previous experiences of inpatient hospitalization especially those experiencing involuntary hospitalization or interactions with law enforcement, described increased adversity during healthcare interactions, as well as diminished trust towards treatment providers, confidence in the benefits of treatment, and engagement in treatment. Furthermore, participants often cited past negative experiences with healthcare as explanations for these outcomes. These results taken together suggest that many young adults referred to EIS, especially those referred from urgent services, are at risk for negative clinical outcomes including relapse which may be influenced by intermediate outcomes such as negative perceptions of EIS and decreased engagement in treatment. As engagement in treatment is associated with improved symptomatic and functional outcomes, this available research highlights the need for additional support to be provided to new patients in EIS in order to address potential negative perceptions towards healthcare and strengthen engagement in treatment which may predict long term clinical outcomes.

A recent trial of a brief engagement intervention called Just Do You, showed promise in addressing barriers to engagement and recovery for young adults with serious mental illness (SMI) and may be useful at the NSEPP. This manualized intervention aimed to strengthen engagement in treatment by facilitating the processing of prior negative experiences with healthcare, empowering participants to take leadership in recovery, thus increasing participants "buy-in" towards treatment. Additionally, the Just Do You intervention was initially designed to be 2 sessions in length. While more intensive psychotherapeutic interventions may provide additional benefit, these are often more resource intensive and associated with increased difficulty with recruitment and maintaining participant engagement. Considering these challenges, a briefer intervention focused on bolstering engagement may be more feasible and cost-effective for a wider population.

Despite the promising results of this initial trial and potential utility of this intervention, key differences between the NSEPP and the services where Just Do You was implemented may detract from the suitability of this intervention in its current form. Firstly, this project was conducted in a different treatment setting (New York) and in a general young adult psychiatric sample (which included but was not exclusive to those experiencing early phase psychosis), who were likely to have less severe illness on average and differing treatment needs compared to an early phase psychosis population. In addition, as a facilitator of engagement during sessions, the Just Do You intervention incorporated elements of music and art therapy modalities. While these appeared efficacious in the initial study, art and music therapy are specialized modalities that most settings (including the NSEPP) do not have resources or expertise to properly implement. As a result, the suitability/feasibility of this intervention for early psychosis populations (young adults) in Canada/Nova Scotia is unclear. This project aims to implement an adapted version of the Just Do You intervention at the NSEPP, to strengthen engagement in treatment for recent referrals.

Study Objectives

In fulfillment of these aims, this project has 6 associated objectives described below:

Primary Objectives Objective 1: Engage patient partners in adapting the Just Do You intervention to ensure its suitability and successful delivery at the NSEPP.

Objective 2: Deliver tailored engagement intervention to recently accepted patients at the NSEPP.

Objective 3: Evaluate the effectiveness of this intervention at improving patient reported measures of treatment engagement, recovery, and insight.

Secondary Objectives

Objective 4: Explore trends in participants' administrative health outcomes as a consequence of intervention, including number of missed appointments, emergency room visits, and hospitalization for psychosis relapse.

Objective 5: Compare trends in administrative outcomes following intervention for patients referred to EIS from urgent services to those referred to EIS from all other sources.

Hypotheses

Based on past research conducted by at the Nova Scotia Early Psychosis Program and results from evaluations of the Just Do You intervention, The investigators hypothesize that for participants in the treatment group, this intervention will lead to i) significant improvement in treatment engagement and recovery over the 3-month follow-up period. Furthermore, the investigators hypothesize that participation in the brief intervention will lead to significantly greater decreases in internalized stigma compared to non-participation over follow-up. Additionally, over 6 months from admission to EIS, it is hypothesized that participants who receive the intervention will display: iii) reduction in missed appointments iv) reduction in number of emergency room visits, and inpatient hospitalizations and v) greater improvements in engagement, recovery, and health outcomes, as measured by effect size, for those referred to EIS from urgent services compared to referrals from other sources following a sub-group analysis.

Participant selection

All participants will be individuals aged 19 to 35 years old who are receiving services at NSEPP located at the Abbie J. Lane hospital, QEII Health Sciences Centre. All participants will have a diagnosis of a psychotic disorder using the DSM-5 criteria for schizophrenia spectrum and other psychotic disorders (e.g., schizophrenia, schizoaffective disorder, schizophreniform disorder, unspecified schizophrenia spectrum and other psychotic disorder, etc. Psychotic disorders must have been diagnosed in the last 5 years to be eligible to receive services at NSEPP; only those who have been accepted to NSEPP will be recruited.

For the current study, participants will be recruited within the first 3-12 months of treatment at the NSEPP. The Just Do You engagement intervention was initially designed to be delivered within the first 4-weeks of participants' treatment in order to maximize the potential long-term benefits of participants' strengthened engagement in treatment. However, concerns have been raised that recruitment within the first four weeks of treatment at NSEPP may not be feasible with an early phase psychosis population who are likely to be experiencing more severe illness compared to those in the original Just Do You trial. As a result, the proposed recruitment timeline was determined in order to ensure recruitment procedures of the current study are as similar to those of the initial Just Do You intervention as is feasible. While this recruitment timeline differs slightly from that of the original Just Do You trial, results from this study support potential benefit of the engagement intervention when delivered after the initial 4-weeks of treatment. Indeed, authors reported that participants who received this intervention after the initial period (50% of overall sample) showed no differences in improvement on outcomes compared to those who received the intervention prior. As a result, it was argued that this intervention may provide benefit even when delivered at various times in participants' treatment.

The investigators will be limiting study participation to those who are aged 19-35. Most early psychosis programs across the country have an age cap of 35 years old, so this restriction is in line with current clinical practices. The investigators aim to recruit 40 participants (20 controls and 20 intervention participants) into the study. The investigators do not anticipate any difficulties with this recruitment strategy as there are currently over 250 active patients at the NSEPP and the program accepts 50-70 new patients to the program each year. The principal investigator, a PhD student in clinical psychology, or a research assistant, will contact the potential participants via telephone, or in person at the NSEPP to provide information about the study at that time, and determine whether participants meet criteria for participation.

Research Plan

Objective 1: Engaging patient partners in adapting the Just Do You intervention.

The initial phase of this project involves active collaboration with patient partners in adapting the Just Do You intervention for suitable use in an early phase psychosis sample. Adaptation of the existing intervention (e.g., choosing suitable resources/exercises to facilitate discussion around past treatment experiences) will involve round table collaborative discussions with study personnel, including the peer support worker, and two members of the EPINS First Voice Advisory Group. Discussions will first be centered around highlighting specific components of the initial Just Do You intervention and discussing intervention acceptability and feasibility of delivery. As concerns may arise, patient partners and study personnel will work collaboratively to modify intervention components to support intervention acceptability while ensuring modifications are consistent with theoretical and empirical underpinnings of the intervention. During initial adaptation stages, emphasis will be placed on actively engaging members of the EPINS First Voice Advisory Group who have had negative experiences with healthcare prior to engaging in EIS to ensure participants' concerns are considered when adapting the Just Do You intervention. It is anticipated that initial intervention adaptation will require a 9-12-hour commitment of each representative over 3, 3- 4-hour initial meetings.

Following adaptation of the intervention, eligible clinicians and the peer support worker will be trained on delivering the intervention by a clinical psychology Ph.D. student, and a licensed clinical psychologist, both of whom have experience working with this population and will be involved in initial adaptation of the Just Do You intervention. Training will involve a full-day workshop lead by investigators which will include presentation of the intervention, treatment targets, underlying theory, and role-play in delivering the intervention with clinicians and PSW. Following training, the investigators will begin delivery of the modified version of the Just Do You intervention to patients at the NSEPP.

During implementation and delivery phase of the project, study personnel will continue to meet with patient representatives once every two months at project steering committee meetings. In these meetings patient representatives will be informed of any study updates and will collaborate with study investigators in finding solutions to encountered challenges including difficulties with intervention delivery or study recruitment. Additionally, when applicable, in steering committee meetings, patient partners and co-investigators will collaborate on reviewing and preparing relevant study material including ethics amendments, consent forms, and materials summarizing study findings to be shared with a broader audience. As this project is anticipated to take 2-years to complete, patient representatives will be required to attend 12, 1-hour meetings with investigators in addition to the initial intervention adaptation meetings.

Throughout patient engagement activities in this project, The Public and Patient Engagement Evaluation Tool (PPEET) will be administered regularly (once after each meeting) to allow patient partners to provide regular feedback to research staff. The PPEET is an evidence-based brief survey measure designed to gain patient partners' assessments of engagement activities throughout the project. Results from this measure will allow investigators to assess degree to which patient partners believe meaningful engagement in project processes has been achieved and results will be used on an ongoing basis to improve engagement processes during the study.

Objective's 2 and 3: Delivering and evaluating the engagement intervention.

Following adaptation of Just Do You, delivery and evaluation of the intervention will begin. A repeated measures quasi-experimental design will be used to evaluate the engagement intervention's effectiveness. This design is most suitable as randomization of participants to treatment or control may be unethical given existing evidence supporting the intervention's effectiveness. Consequently, the investigators aim to approach all eligible patients within the first 3-12 months of treatment who have previously consented to being contacted for research purposes (roughly 80% of overall patient population). Eligible patients will be informed of the study protocol/rationale, as well as potential risks and benefits of participation in the intervention. Following this, eligible participants will choose between i) full participation in the treatment group, which involves engaging in the 2-part treatment intervention and completing study outcome assessments ii) participation in the control group which involves completing outcome assessments during regular clinical visits without engaging in the intervention and iii) refraining from participating in the study. Following this, those expressing interest in participating in either the treatment or control conditions will engage in a more in-depth consent discussion where additional specifics of participation will be outlined including risks/benefits, confidentiality, and the study protocol. Individuals providing informed consent to participate in the study will then complete a baseline assessment. This assessment includes completion of a demographic form which will include questions about participants' age, ethnicity, migrant status, gender identity, and sexual orientation , as well as questions about participants' past experiences with mental healthcare and referral source. In addition, participants postal code will be collected and used to extrapolate an estimate of participants' socioeconomic status (SES) using The Canadian Index of Multiple Deprivation (CIMD). This index developed by Statistics Canada, uses postal code data to estimate individuals' SES using participants' geographical location on four dimensions: Residential instability, Economic dependency, Ethno-cultural composition, and Situational vulnerability. These dimensions based on available evidence and up-to date census data, and are widely used in Canadian health research as proxy multi-dimensional estimates of SES. Collection of demographic data will allow investigators to better describe the participant sample and potentially allow for exploration of potential differential outcomes in minority communities.

Participants will then complete a baseline clinical assessment which includes measures of engagement in treatment (Yatchmenoff Client Engagement Scale), self-reported recovery (Recovery Assessment Scale), psychotic symptom severity (PANSS-6), global impression of illness severity Clinical (CGI-I and -S) Social and Occupational Functioning (SOFAS), illness insight (SUMD), current substance use (WHO-ASSIST FC), experiences of adverse and traumatic life events (TALE), and self/internalized stigma (ISMI). These measures have all been validated and previously used in early psychosis populations. The engagement and recovery measures were previously employed by investigators in the initial Just Do You trial and have been chosen to ensure comparability between studies.

Intervention Procedure and Follow-up

Following baseline assessment, participants receiving the intervention will engage in two intervention modules (between 90-120 minutes each) led by a clinician and PSW. This intervention is based on the "young adult framework" for mental health and is informed by theories of health behaviour change and formal decision theory. Targets of these sessions are common cognitive and affective barriers to engagement in mental health services for young adults, especially those with past negative experiences with healthcare (e.g., behavioural beliefs, image impressions, emotional reactions, personal efficacy, norms). Following outlined practices, and to reduce burden of participation, participants will engage in the first module immediately following baseline assessment. Module 1 will focus on discussions of the recovery process and principles of recovery while exploring stigma and participants' perceptions and attitudes towards clinical service. Module 2 , which will be delivered 4-weeks following the first session, will focus on processing prior difficult experiences with healthcare and psychosis, and resulting perceptions towards treatment that commonly act as barriers to engagement. Emphasis will be placed on instilling participants hope in recovery and building trust in current EIS.

As the NSEPP largely provides care in person, and study sessions are designed to coincide with participants regular treatment sessions at NSEPP, Participants will be encouraged to complete the intervention modules in person. However, in order to increase accessibility to the intervention for participants who may have increased difficulty travelling to NSEPP, participants will be given the option to attend sessions virtually through Zoom for Healthcare. This interface has been carefully vetted by NS health for use with patients and is deemed to be the most secure virtual method to ensure patient/participant privacy and security. In addition to a baseline assessment, treatment and control groups will complete follow up measures of participants' self reported recovery and engagement outcomes 2 and 4-weeks following initial study enrollment. Finally, participants in the treatment group will complete assessment measures 3-months post-delivery of second session, and control participants will complete measures 4-months following enrollment. At final assessment, participants' PANSS-6, CGI-I, SOFAS, SUMD, WHO-ASSIST and ISMI-9 scores will be measured in addition to participants' recovery (RAS), and engagement scores (Yatchmenoff client engagement scale). Based on preference, participants will be provided the option to complete self report measures at follow-up times either in person at the NSEPP, or virtually. Those electing to complete follow-up measures through REDCap, will be invited by email to complete the web-based self-report measures. De-identified data will be automatically entered into the secure web-based REDCap database capture platform with only participant ID approved by NS Health and managed in accordance with provincial privacy standards. For participants electing to complete measures virtually, clinician rated assessments will be completed in person at the NSEPP or completed virtually via Zoom for healthcare for NSHealth. Completion of the above protocol will translate to a total length of follow up of 4 months for all participants

Objective's 4 and 5: Monitoring administrative health outcomes:

In addition to evaluating effectiveness of the intervention by administering the above outcomes, administrative health data will be used to explore intervention impact on participants high level clinical outcomes. Firstly, to obtain an additional objective indicator of participants' treatment engagement, the investigators will measure participants' rate of missed appointments 3-months prior and 6-months following intervention. In addition, the investigators will measure rate of hospitalization and ER visits over the same time (cumulative # of visits/person-year). As the investigators have prior ethics approval to monitor high level demographic and outcome data for all NSEPP patients (including those accepted to treatment who never engaged in EIS), the investigators will use all past and present patients who did not receive the intervention as a comparison group and measure participants' administrative health outcomes over the same timeline. Finally, outcomes for participants referred to NSEPP from urgent services will be compared to those of participants referred from other services to assess differential effectiveness of the intervention in previously identified high-risk groups.

Data analysis plan

The goal of this project is to adapt the Just Do You intervention for use at NSEPP and deliver and evaluate the effectiveness of this intervention. In accordance with the stated objectives and consistent with the initial Just Do You trial, the investigators will measure changes in participants' engagement, recovery, insight, stigma and symptoms over follow-up and compare changes on these outcomes between control and active participants. To address this first hypothesis - that participants who engaged in the intervention will show greater improvements in engagement, self-reported recovery, and insight, compared to those in the control condition, the investigators will use linear mixed regression models which are most suitable for repeated measures designs. Potential differences in overall illness severity (CGI-S, PANSS-6, SOFAS, WHO-ASSIST) between control and treatment groups at baseline will be assessed using independent t-tests. If significant differences on these measures are observed between groups, baseline scores on these outcomes will be included as predictors in analyses, in addition to treatment group. The investigators aim to recruit 40 participants (20 controls and 20 intervention participants) into the study. This sample size was calculated to ensure 80% power of detecting the minimum effect size previously reported in the trial of the Just Do You intervention (Cohen's D ranged from 0.50 to 1.15). This sample is feasible given the clinic's large patient pool (250+ active patients, 50 -70 new admissions/year) and the nature of research at NSEPP being embedded into clinical practice. To measure impact of the intervention on participants' self reported engagement, recovery, and insight, the investigators will use linear mixed regression models which are suitable for repeated measures designs.

To address the second and third hypotheses (in fulfillment of study objectives 4 and 5) - that those receiving the study intervention will show a trend of fewer overall emergency department visits and hospitalizations for mental health reasons, as well as fewer missed treatment appointments compared to those who received treatment as usual, Poisson regression models will be used. To assess for trends in rate of missed appointments, hospitalization, and ER visits and to compare potential differential outcomes for those referred to EIS via urgent or non-urgent sources, both treatment group and referral source (i.e., urgent vs non-urgent referral will be included as predictors in analyses using time of follow up as an offset variable in analysis. If after reviewing the distribution of hospitalizations, Poisson regression does not fit the data well, (i.e., data are over dispersed or are characterized by considerable proportion of sample not having urgent care visits) modified Poisson regression can be used: If the sample variance is significantly greater than the mean number of outcomes, negative binomial regression will be used to account for this extra variance. If data are skewed towards zero hospitalizations, A zero inflated Poisson model will be used.

Due to the small sample size (20 active participants and 20 controls, with potential to include roughly 500 additional retrospective controls) the investigators may not be adequately powered to detect small differences in administrative health outcomes between participant groups or include additional important demographic and clinical variables in analyses. Nonetheless, as this is a pilot project, the investigators will assess and to report observed trends in health outcomes which are anticipated to act as preliminary "proof of concept" findings supporting potential subsequent follow-up studies. It is the investigators aim that these initial study findings will facilitate potential follow-up studies evaluating this intervention that are adequately powered to detect differences in administrative health outcomes while control for additional potential confounders.

To address the fourth hypothesis - That participant's with past urgent service referral will benefit more from the intervention than those referred from other sources (e.g., GP, family/self Community mental health), Subgroup comparisons will be conducted. The overall effect size, attributable to the intervention, measured with Cohen's D, will be compared between participants with urgent vs non urgent referral to EIS.

Confidentiality

The principal investigator will keep a file that links participant ID numbers to names that will be password-protected and stored on a computer that is housed at the Abbie J Lane building. The only location where identifying information will be kept will be on the secure computer at NSEPP; this information will be kept in a password-protected file and will be accessible only to the principal investigator, and supervising investigators, if necessary; Research assistants and the peer support worker will have access to the de-identified file that contains ID numbers and the remainder of participant information (e.g., outcomes). In addition to being in a locked room in the NSEPP. The computer on which files will be stored is also encrypted, to prevent a breach of confidentiality should the computer be lost or stolen. Potential participants' contact information and information regarding date of acceptance to the NSEPP will be taken from the NSEPP clinic database of those participants who gave prior consent to the clinic to release this information for research purposes, limiting the need to gain access to the potential participant's health record. Completed measures, either paper and pencil or virtually through REDCap will be stored only with the date and unique participant ID number; names or other identifying information will not be used. Paper questionnaires will be kept separately each in a separate locked filing cabinet in a locked room with limited access. Participant ID number and identifying information will be linked only through the password-protected file located on the principal investigator's computer housed at the NSEPP. Consent forms will be stored under lock and key in the principal investigator's office at Abbie J Lane, as will study data (stored in a separate locked filing cabinet). Seven years following the publication of the study results, all data will be destroyed/permanently erased, as required by the Nova Scotia Health Authority. The records on the principal investigator's computer will be permanently erased by the principal investigator with the assistance of IT, and the physical records at the Abbie J Lane hospital will also be destroyed by the PI.

ELIGIBILITY:
Inclusion Criteria:

* Within first 3-12 months of treatment in early intervention services.
* Diagnosis of a psychotic disorder using the DSM-5 criteria for schizophrenia spectrum and other psychotic disorders (e.g., schizophrenia, schizoaffective disorder, schizophreniform disorder, unspecified schizophrenia spectrum and other psychotic disorder, etc.)
* Diagnosis within past 5 years.

Exclusion Criteria:

* Primary diagnosis that is not a psychotic disorder.
* Outside of age limits.
* Intellectual Disability (IQ < 70)

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Yatchmenoff Client Engagement Scale - Modified | Administered at baseline (T0), 2 weeks follow up, 4 weeks follow-up and at end of study follow up at 4 months.
  Participants' self-reported engagement in treatment is measured using a modified version of the Yatchmenoff Client Engagement Scale. Initially designed to assess engagement in child protective services, but previously modified and used in the initial Just Do You trial, modification of this scale will involve for this study slight changes to wording of questions to different care setting. This 19-item measure assesses respondents' perceptions of treatment and engagement in it across 4 dimensions using a 5-point likert scale with responses ranging from 1 - Strongly Disagree to 5 - Strongly Agree: Receptivity (Range: 4 - 20, with higher scores indicating increased receptivity to treatment) Buy-in (Range: 8 - 40, with higher scores indicating increased buy-in to treatment), Working relationship (Range: 4 - 20, with higher scores indicating perceptions of a stronger working relationship), and Trust (Range: 3 - 15, with higher scores indicating increased trust in care providers).
Recovery Assessment Scale - Revised (RAS-R) | Administered at baseline (T0), 2-weeks follow up, 4 weeks follow-up and at end of study follow up at 4 months.
  Participants' recovery is measured using the 24-item revised version of the Recovery Assessment Scale (RAS-R). The RAS is a self-report assessment of individuals' recovery, previously determined to be valid for use with those experiencing serious mental illness. The RAS-R assesses respondents' perceptions of personal recovery in 5 domains: Personal confidence and hope, Willingness to ask for help, Goal and success orientation, Reliance on others, and No domination by symptoms. Responses are scored using a 5-point likert scale with responses ranging from 1 - Strongly Disagree to 5 - Strongly Agree. Total scores range from 24 - 120 with higher values indicating respondents' perceptions of more improved recovery.
9-item Internalized Stigma of Mental Illness Inventory (ISMI-9) | Administered at baseline (T0) and at end of study follow up at 4 months.
  Participants' internalized stigma will be measured using the abbreviated 9-item Internalized Stigma of Mental Illness Inventory (ISMI-9). The ISMI-9 is an abbreviated version of the original 29 item ISMI, that aims to assess degree of internalized/self stigma in those experiencing mental illness. Each item of the scale is measured on a 4-point Likert scale (1 - strongly disagree to 4 - strongly agree). Total are then divided by 9 to obtain an average score for internalized stigma with higher scores indicating greater degrees of internalized stigma for respondents (Range: 1 - 4). The 29-item version of this scale has been widely used in studies of stigma in early psychosis samples, but the abbreviated version will be used for this study to reduce burden of involvement on study participants. The 9-item version has been previously demonstrated to have adequate psychometric properties.

SECONDARY OUTCOMES:
Positive and Negative Syndrome Scale 6-item abbreviated version (PANSS-6) | Administered at baseline (T0) and at end of study follow up at 4 months.
  Psychotic symptoms are measured using the Positive and Negative Syndrome Scale 6-item abbreviated version, a validated abbreviated version of the PANSS-30 gold standard measure of symptom severity in psychosis. This clinician-rated measure assesses respondents' symptom severity using 6-items from the original 30 item PANSS (P1-Delusions, P2-Conceptual disorganization, P3- Hallucinations, N1- Blunted affect, N4- Social withdrawal, N6 - Lack of spontaneity and flow of conversation). Item scores range from 1 - minimal symptoms to 7 - extreme symptoms with increased PANSS-6 total scores indicating more severe symptoms (Range: 6 - 42).
Clinical Global Impression (CGI-I & CGI-S) | Administered at baseline (T0) and at end of study follow up at 4 months.
  Assessment of participants global illness severity will be assessed using the CGI-S. The CGI-S is a 7-point clinician rated Likert scale that assesses individuals' overall illness severity relative those who the clinician has experienced with the same diagnosis (ranging from 1 = Normal, not at all ill to 7 = Extremely ill). The CGI-I is a 7-point clinician rated Likert scale that assesses an individual's global change in illness severity compared to a baseline rating prior to intervention (ranging from 1 = Very much improved to 7 = Very much worse).
Social and Occupational Functioning Assessment Scale (SOFAS) | Administered at baseline (T0) and at end of study follow up at 4 months.
  Functioning is measured using the Social and Occupational Functioning Assessment Scale (SOFAS). The SOFAS is a widely used, reliable, clinician determined, single item measure of individuals' social and occupational functioning independent of symptoms. The SOFAS is a 100-point single-item rating measure, subdivided into 10 equal intervals (Range: 0 - 100) with higher scores indicating improved functioning.
Abbreviated Scale to Assess Unawareness in Mental Disorder (SUMD) | Administered at baseline (T0) and at end of study follow up at 4 months.
  Participant insight will be measured using the Abbreviated Scale to Assess Unawareness in Mental Disorder (SUMD). This is a 9-item clinician administered measure of participants' insight which is commonly impaired in psychosis. The SUMD assesses insight along 3 core dimensions determined to: Awareness of the disease, Consequences and need for treatment; Awareness of symptoms. The scores are typically measured on a scale from 0 to 100, with higher scores indicating better insight.
WHO Alcohol, Smoking, and Substance Involvement Screening Test (ASSIST) - FC | Administered at baseline (T0) and at end of study follow up at 4 months.
  Participant substance use will be measured using A modified version of the WHO Alcohol, Smoking, and Substance Involvement Screening Test (ASSIST), called the ASSIST-FC. This measure asks participants about frequency of use and potential for misuse using two questions: "In the past 3 months, which of the following substances have you used?", "Has a friend or relative or anyone else ever expressed concern about your use of any substances?"). Possible answers range from "Never" to "Daily or almost daily" for the first question and for the second question, range from "No, never", "Yes, in the past 3 months," to "Yes, but not in the past 3 months." The full ASSIST is regularly used at the Nova Scotia Early Psychosis Program (NSEPP), but the shortened version will be used to decrease burden of study involvement for participants.
The Trauma and Life Events (TALE) checklist | Administered at baseline (T0)
  Experiences of Traumatic/Adverse Events Participants' experiences of lifetime traumatic events will be measured using The Trauma and Life Events (TALE) checklist. The TALE is a 21-item questionnaire, which assesses what adverse experiences participants have experienced, when they happened and the number of experiences of these events. Additionally, this questionnaire assesses the degree to which endorsed adverse events are affecting participants now in any way.
Demographic Questionnaire | Administered at baseline (T0)
  Participants' demographic characteristics will be assessed using a demographic form which will include questions about participants' age, ethnicity, migrant status, gender identity, and sexual orientation, as well as questions about past experiences with mental healthcare and referral source. In addition, participants postal code will be collected and used to extrapolate an estimate of socioeconomic status (SES) using The Canadian Index of Multiple Deprivation (CIMD). This index developed by Statistics Canada, uses postal code data to estimate individuals' SES using participants' geographical location on four dimensions: Residential instability, Economic dependency, Ethno-cultural composition, and Situational vulnerability. These dimensions based on available evidence and up-to date census data, and are widely used in Canadian health research as proxy multi-dimensional estimates of SES.

OTHER OUTCOMES:
Quantitative Engagement: Rate of Missed Appointments | Number/rate of missed appointments will begin being measured 3-month's prior to involvement in the study and end 6-months following initial engagement in the study.
  In order to obtain an additional objective indicator of participants' treatment engagement, we will measure participants' rate of missed appointments 3-months prior and 6-months following intervention. Number of missed appointments will be compared for treatment vs control participants to assess whether the treatment intervention is associated with a reduction in missed appointments.
Rate of Emergency Department Visits & Hospital Admissions | Number/rate of missed appointments will begin being measured 3-month's prior to involvement in the study and end 6-months following initial engagement in the study.
  In addition, we will measure rate of hospitalization and ER visits (cumulative # of visits/person-month) over the same time frame (3-months prior and 6-months following intervention). Rate of ER and hospital admissions will be compared for treatment vs control participants to assess whether the treatment intervention is associated with a difference in urgent service use between the treatment and control group.

CONTACTS AND LOCATIONS:
Overall Officials: Phil Tibbo, MD, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Nova Scotia Early Psychosis Program (NSEPP), Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: Yes
In order to ensure privacy of other participants is respected we will not be making data available to other researchers unless it is requested and sharing has been approved by our institution.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Following study completion and result publication in roughly Spring 2027
Access Criteria: Available upon request with information to contact provided in published manuscript.

REFERENCES:
- [Background] Bertolote J, McGorry P. Early intervention and recovery for young people with early psychosis: consensus statement. Br J Psychiatry Suppl. 2005 Aug;48:s116-9. doi: 10.1192/bjp.187.48.s116. PMID 16055800
- [Background] Addington J, Van Mastrigt S, Hutchinson J, Addington D. Pathways to care: help seeking behaviour in first episode psychosis. Acta Psychiatr Scand. 2002 Nov;106(5):358-64. doi: 10.1034/j.1600-0447.2002.02004.x. PMID 12366470
- [Background] Weiss A, Steadman S, Mercier HD, Hansel TC, Chaudhry S, Clark I. Pathways to Care: How Help-Seeking Behaviors Relate to Duration of Untreated Psychosis and Treatment Engagement. Psychiatr Q. 2022 Jun;93(2):473-482. doi: 10.1007/s11126-021-09960-5. Epub 2021 Oct 20. PMID 34669120
- [Background] Jones N, Gius BK, Shields M, Collings S, Rosen C, Munson M. Investigating the impact of involuntary psychiatric hospitalization on youth and young adult trust and help-seeking in pathways to care. Soc Psychiatry Psychiatr Epidemiol. 2021 Nov;56(11):2017-2027. doi: 10.1007/s00127-021-02048-2. Epub 2021 Mar 9. PMID 33751175
- [Background] Anderson KK, Fuhrer R, Schmitz N, Malla AK. Determinants of negative pathways to care and their impact on service disengagement in first-episode psychosis. Soc Psychiatry Psychiatr Epidemiol. 2013 Jan;48(1):125-36. doi: 10.1007/s00127-012-0571-0. Epub 2012 Sep 14. PMID 22976337
- [Background] Rodrigues R, Anderson KK. The traumatic experience of first-episode psychosis: A systematic review and meta-analysis. Schizophr Res. 2017 Nov;189:27-36. doi: 10.1016/j.schres.2017.01.045. Epub 2017 Feb 14. PMID 28214175
- [Background] MacDonald K, Fainman-Adelman N, Anderson KK, Iyer SN. Pathways to mental health services for young people: a systematic review. Soc Psychiatry Psychiatr Epidemiol. 2018 Oct;53(10):1005-1038. doi: 10.1007/s00127-018-1578-y. Epub 2018 Aug 22. PMID 30136192
- [Background] Seed T, Fox JR, Berry K. The experience of involuntary detention in acute psychiatric care. A review and synthesis of qualitative studies. Int J Nurs Stud. 2016 Sep;61:82-94. doi: 10.1016/j.ijnurstu.2016.05.014. Epub 2016 Jun 4. PMID 27314181
- [Background] Silva B, Bachelard M, Amoussou JR, Martinez D, Bonalumi C, Bonsack C, Golay P, Morandi S. Feeling coerced during voluntary and involuntary psychiatric hospitalisation: A review and meta-aggregation of qualitative studies. Heliyon. 2023 Feb 2;9(2):e13420. doi: 10.1016/j.heliyon.2023.e13420. eCollection 2023 Feb. PMID 36820044
- [Background] Priebe S, Katsakou C, Amos T, Leese M, Morriss R, Rose D, Wykes T, Yeeles K. Patients' views and readmissions 1 year after involuntary hospitalisation. Br J Psychiatry. 2009 Jan;194(1):49-54. doi: 10.1192/bjp.bp.108.052266. PMID 19118325
- [Background] Priebe S, Katsakou C, Glockner M, Dembinskas A, Fiorillo A, Karastergiou A, Kiejna A, Kjellin L, Nawka P, Onchev G, Raboch J, Schuetzwohl M, Solomon Z, Torres-Gonzalez F, Wang D, Kallert T. Patients' views of involuntary hospital admission after 1 and 3 months: prospective study in 11 European countries. Br J Psychiatry. 2010 Mar;196(3):179-85. doi: 10.1192/bjp.bp.109.068916. PMID 20194537
- [Background] Mueser KT, Lu W, Rosenberg SD, Wolfe R. The trauma of psychosis: posttraumatic stress disorder and recent onset psychosis. Schizophr Res. 2010 Feb;116(2-3):217-27. doi: 10.1016/j.schres.2009.10.025. Epub 2009 Nov 24. PMID 19939633
- [Background] Minsky SK, Lu W, Silverstein SM, Gara M, Gottlieb JD, Mueser KT. Service Use and Self-Reported Symptoms Among Persons With Positive PTSD Screens and Serious Mental Illness. Psychiatr Serv. 2015 Aug 1;66(8):845-50. doi: 10.1176/appi.ps.201400192. Epub 2015 Apr 15. PMID 25873024
- [Background] Senger B, Pencer A, Crocker CE, Simon P, Taylor B, Tibbo PG. The role of referral pathway to early intervention services for psychosis on 2-year inpatient and emergency service use. J Psychiatr Res. 2024 Apr;172:340-344. doi: 10.1016/j.jpsychires.2024.02.035. Epub 2024 Feb 28. PMID 38442449
- [Background] Dixon LB, Holoshitz Y, Nossel I. Treatment engagement of individuals experiencing mental illness: review and update. World Psychiatry. 2016 Feb;15(1):13-20. doi: 10.1002/wps.20306. PMID 26833597
- [Background] Macbeth A, Gumley A, Schwannauer M, Fisher R. Service engagement in first episode psychosis: clinical and premorbid correlates. J Nerv Ment Dis. 2013 May;201(5):359-64. doi: 10.1097/NMD.0b013e31828e0e19. PMID 23588222
- [Background] Munson MR, Jaccard JJ, Scott LD Jr, Narendorf SC, Moore KL, Jenefsky N, Cole A, Davis M, Gilmer T, Shimizu R, Pleines K, Cooper K, Rodwin AH, Hylek L, Amaro A. Engagement intervention versus treatment as usual for young adults with serious mental illness: a randomized pilot trial. Pilot Feasibility Stud. 2020 Jul 23;6:107. doi: 10.1186/s40814-020-00650-w. eCollection 2020. PMID 32714561
- [Background] Munson MR, Jaccard J, Moore KL, Rodwin AH, Shimizu R, Cole AR, Scott LD Jr, Narendorf SC, Davis M, Gilmer T, Stanhope V. Impact of a brief intervention to improve engagement in a recovery program for young adults with serious mental illness. Schizophr Res. 2022 Dec;250:104-111. doi: 10.1016/j.schres.2022.11.008. Epub 2022 Nov 15. PMID 36399899
- [Background] Abelson J, Li K, Wilson G, Shields K, Schneider C, Boesveld S. Supporting quality public and patient engagement in health system organizations: development and usability testing of the Public and Patient Engagement Evaluation Tool. Health Expect. 2016 Aug;19(4):817-27. doi: 10.1111/hex.12378. Epub 2015 Jun 25. PMID 26113295
- [Background] Kontopantelis E, Doran T, Springate DA, Buchan I, Reeves D. Regression based quasi-experimental approach when randomisation is not an option: interrupted time series analysis. BMJ. 2015 Jun 9;350:h2750. doi: 10.1136/bmj.h2750. PMID 26058820
- [Background] Street LL, Luoma JB. Control groups in psychosocial intervention research: ethical and methodological issues. Ethics Behav. 2002;12(1):1-30. doi: 10.1207/S15327019EB1201_1. PMID 12171079
- [Background] Statistics Canada. 2019. "The Canadian Index of Multiple Deprivation". Statistics Canada Catalogue no. 45-20-0001.
- [Background] Matheson FI, Dunn JR, Smith KL, Moineddin R, Glazier RH. Development of the Canadian Marginalization Index: a new tool for the study of inequality. Can J Public Health. 2012 Apr 30;103(8 Suppl 2):S12-6. doi: 10.1007/BF03403823. PMID 23618065
- [Background] D. K. Yatchmenoff, "Measuring client engagement from the client's perspective in nonvoluntary child protective services," Res. Soc. Work Pract., vol. 15, no. 2, pp. 84-96, 2005.
- [Background] Corrigan PW, Salzer M, Ralph RO, Sangster Y, Keck L. Examining the factor structure of the recovery assessment scale. Schizophr Bull. 2004;30(4):1035-41. doi: 10.1093/oxfordjournals.schbul.a007118. PMID 15957202
- [Background] Salzer MS, Brusilovskiy E. Advancing recovery science: reliability and validity properties of the Recovery Assessment Scale. Psychiatr Serv. 2014 Apr 1;65(4):442-53. doi: 10.1176/appi.ps.201300089. PMID 24487405
- [Background] Kaplan K, Salzer MS, Brusilovskiy E. Community participation as a predictor of recovery-oriented outcomes among emerging and mature adults with mental illnesses. Psychiatr Rehabil J. 2012 Winter;35(3):219-29. doi: 10.2975/35.3.2012.219.229. PMID 22246120
- [Background] Kay SR, Fiszbein A, Opler LA. The positive and negative syndrome scale (PANSS) for schizophrenia. Schizophr Bull. 1987;13(2):261-76. doi: 10.1093/schbul/13.2.261. PMID 3616518
- [Background] W. Guy, "Clinical Global Impression," in Assessment manual for psychopharmacology, Rockville, MD: US Department of Health, Education, and Welfare, 1976.
- [Background] Morosini PL, Magliano L, Brambilla L, Ugolini S, Pioli R. Development, reliability and acceptability of a new version of the DSM-IV Social and Occupational Functioning Assessment Scale (SOFAS) to assess routine social functioning. Acta Psychiatr Scand. 2000 Apr;101(4):323-9. PMID 10782554
- [Background] Amador XF, Strauss DH, Yale SA, Flaum MM, Endicott J, Gorman JM. Assessment of insight in psychosis. Am J Psychiatry. 1993 Jun;150(6):873-9. doi: 10.1176/ajp.150.6.873. PMID 8494061
- [Background] Michel P, Baumstarck K, Auquier P, Amador X, Dumas R, Fernandez J, Lancon C, Boyer L. Psychometric properties of the abbreviated version of the Scale to Assess Unawareness in Mental Disorder in schizophrenia. BMC Psychiatry. 2013 Sep 22;13:229. doi: 10.1186/1471-244X-13-229. PMID 24053640
- [Background] WHO ASSIST Working Group. The Alcohol, Smoking and Substance Involvement Screening Test (ASSIST): development, reliability and feasibility. Addiction. 2002 Sep;97(9):1183-94. doi: 10.1046/j.1360-0443.2002.00185.x. PMID 12199834
- [Background] McRee B, Babor TF, Lynch ML, Vendetti JA. Reliability and Validity of a Two-Question Version of the World Health Organization's Alcohol, Smoking and Substance Involvement Screening Test: The ASSIST-FC. J Stud Alcohol Drugs. 2018 Jul;79(4):649-657. PMID 30079882
- [Background] Carr S, Hardy A, Fornells-Ambrojo M. The Trauma and Life Events (TALE) checklist: development of a tool for improving routine screening in people with psychosis. Eur J Psychotraumatol. 2018 Sep 11;9(1):1512265. doi: 10.1080/20008198.2018.1512265. eCollection 2018. PMID 30220986
- [Background] Hammer, J. H., & Toland, M. D. (2017). Internal structure and reliability of the Internalized Stigma of Mental Illness Scale (ISMI-29) and Brief Versions (ISMI-10, ISMI-9) among Americans with depression. Stigma and Health, 2(3), 159.
- [Background] Boyd JE, Adler EP, Otilingam PG, Peters T. Internalized Stigma of Mental Illness (ISMI) scale: a multinational review. Compr Psychiatry. 2014 Jan;55(1):221-31. doi: 10.1016/j.comppsych.2013.06.005. Epub 2013 Sep 21. PMID 24060237
- [Background] West BT. Analyzing longitudinal data with the linear mixed models procedure in SPSS. Eval Health Prof. 2009 Sep;32(3):207-28. doi: 10.1177/0163278709338554. Epub 2009 Aug 13. PMID 19679634
- [Background] Liu S, Rovine MJ, Molenaar PC. Selecting a linear mixed model for longitudinal data: repeated measures analysis of variance, covariance pattern model, and growth curve approaches. Psychol Methods. 2012 Mar;17(1):15-30. doi: 10.1037/a0026971. Epub 2012 Jan 16. PMID 22251268
- [Background] Weaver CG, Ravani P, Oliver MJ, Austin PC, Quinn RR. Analyzing hospitalization data: potential limitations of Poisson regression. Nephrol Dial Transplant. 2015 Aug;30(8):1244-9. doi: 10.1093/ndt/gfv071. Epub 2015 Mar 25. PMID 25813274
- [Background] Becker-Blease KA, Freyd JJ. Research participants telling the truth about their lives: the ethics of asking and not asking about abuse. Am Psychol. 2006 Apr;61(3):218-26. doi: 10.1037/0003-066X.61.3.218. PMID 16594838